CLINICAL TRIAL: NCT03554291
Title: Repurposing a Histamine Antagonist to Benefit Patients With Pulmonary Hypertension
Acronym: REHAB-PH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Peter Leary, Director, Pulmonary Vascular Disease Program, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005002; 1R61HL142539-01 (NIH)
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Arterial Hypertension; Right Heart Failure
Keywords: famotidine; H2 blocker; H2 antagonist
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Failure | interventions — Famotidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Famotidine (Experimental): 20mg of oral famotidine (pill) daily
  Other names: Pepcid
  Interventions: Drug: Famotidine 20 MG
- Placebo (Placebo Comparator): Daily oral placebo (pill)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Famotidine 20 MG — Famotidine 20 mg capsule taken daily for 24 weeks.
  Arms: Famotidine
Other: Placebo — Placebo capsule taken daily for 24 weeks.
  Arms: Placebo

SUMMARY:
This is a Phase 2, single-center, randomized placebo controlled trial of famotidine (an H2 receptor antagonist) in adults with pulmonary arterial hypertension. The study will evaluate the safety and clinical efficacy of a 24-week course of famotidine.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is one of many conditions that put stress and strain on the right side of the heart. This stress and strain can cause right heart failure. Although there are medications to treat PAH, there are currently no medications that act directly on the heart to improve right heart function. This is different than left heart failure where one of the cornerstones of treatment is medication targeted at the heart to improve left heart function.

Famotidine is a well-tolerated, over-the-counter, and inexpensive medication. Preliminary results suggest that famotidine may help the right heart to adapt and strengthen when stressed instead of fail; however, these results are suggestive and not definitive. A randomized controlled trial is required to evaluate the possibility that famotidine can impact right heart function.

Participants in the study will take famotidine or placebo for 24 weeks. They will have three study visits at 0, 12, and 24 weeks. These visits will add 20-30 minutes to the standard clinic visits at those time points and there will be an echocardiogram at weeks 0 and 24. There will also be one phone visit at 4 weeks to check-in. Some participants may elect to participate in exercise testing and/or right heart catheterization at weeks 0 and 24; however, this is not required to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 80
* WHO Group 1 Pulmonary Arterial Hypertension
* NYHA Functional Class II, III, or IV at screening
* Stable dose of pulmonary vasodilators for 30 days prior to randomization
* Right heart catheterization within five years demonstrating a mean pulmonary arterial pressure of ≥ 25 mmHg, occlusion pressure of ≤ 15 mmHg, and pulmonary vascular resistance of ≥ 3 wood units
* Participants with a right heart catheterization within five years demonstrating a mean pulmonary arterial pressure of ≥ 25 mmHg and occlusion pressure of 15 - 20 mmHg will be considered for inclusion if the pulmonary vascular resistance ≥ 9 wood units and they are being treated with pulmonary arterial hypertension specific therapy
* Able to walk with/without a walking aid for a distance of at least 50 meters

Exclusion Criteria:

* Pregnant or lactating
* Non-group 1 pulmonary hypertension or veno-occlusive disease
* History of interstitial lung disease, unless subject has collagen vascular disease and has pulmonary function testing conducted within 12 months demonstrating a total lung capacity of ≥ 60 %
* Has received or will receive an investigational drug, device, or study within 30 days or during the course of study
* Left sided myocardial disease as evidenced by left ventricular ejection fraction < 40%
* Any other clinically significant illness or abnormal laboratory values (measured during the Screening period) that, in the opinion of the Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data
* Anticipated survival less than 1 year due to concomitant disease
* Regularly taking an H2 receptor antagonist within 30 days of enrollment
* Creatinine clearance < 30 mL/min
* History of bariatric surgery
* Current treatment for HIV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Leary, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leary PJ, Barr RG, Bluemke DA, Bristow MR, Kronmal RA, Lima JA, Ralph DD, Ventetuolo CE, Kawut SM. H2 receptor antagonists and right ventricular morphology: the MESA right ventricle study. Ann Am Thorac Soc. 2014 Nov;11(9):1379-86. doi: 10.1513/AnnalsATS.201407-344OC. PMID 25295642
- [Background] Leary PJ, Tedford RJ, Bluemke DA, Bristow MR, Heckbert SR, Kawut SM, Krieger EV, Lima JA, Masri CS, Ralph DD, Shea S, Weiss NS, Kronmal RA. Histamine H2 Receptor Antagonists, Left Ventricular Morphology, and Heart Failure Risk: The MESA Study. J Am Coll Cardiol. 2016 Apr 5;67(13):1544-1552. doi: 10.1016/j.jacc.2016.01.045. PMID 27150686
- [Background] Leary PJ, Kronmal RA, Bluemke DA, Buttrick PM, Jones KL, Kao DP, Kawut SM, Krieger EV, Lima JA, Minobe W, Ralph DD, Tedford RJ, Weiss NS, Bristow MR. Histamine H2 Receptor Polymorphisms, Myocardial Transcripts, and Heart Failure (from the Multi-Ethnic Study of Atherosclerosis and Beta-Blocker Effect on Remodeling and Gene Expression Trial). Am J Cardiol. 2018 Jan 15;121(2):256-261. doi: 10.1016/j.amjcard.2017.10.016. Epub 2017 Oct 20. PMID 29191567
- [Background] Leary PJ, Hess E, Baron AE, Branch KR, Choudhary G, Hough CL, Maron BA, Ralph DD, Ryan JJ, Tedford RJ, Weiss NS, Zamanian RT, Lahm T. H2 Receptor Antagonist Use and Mortality in Pulmonary Hypertension: Insight from the VA-CART Program. Am J Respir Crit Care Med. 2018 Jun 15;197(12):1638-1641. doi: 10.1164/rccm.201801-0048LE. No abstract available. PMID 29437490
- [Derived] Leary PJ, Rayner SG, Branch KRH, Hogl L, Liston NM, Barros LM, Prout J, Nolley S, Buber J, Ralph DD, Probstfield JL. Effect of Famotidine on Outcomes in Pulmonary Arterial Hypertension: A Randomized Controlled Trial. Chest. 2025 Jul;168(1):189-199. doi: 10.1016/j.chest.2024.12.029. Epub 2025 Jan 4. PMID 39761829

RESULTS

PARTICIPANT FLOW:
Groups:
- Famotidine: 20mg of oral famotidine (pill) daily
  Other names: Pepcid
  Famotidine 20 MG: Famotidine 20 mg capsule taken daily for 24 weeks.
Period: Overall Study
Arm/Group | Famotidine | Placebo
Started | 41 | 39
Completed | 34 | 38
Not Completed | 7 | 1
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — COVID Travel Restriction- Partial Data Collected | 3 | 0

BASELINE CHARACTERISTICS:
Population: One participant withdrew from the study after randomization but before receipt of study drug and without knowledge of their assigned arm. They were not included in analyses in accordance with the plan to proceed with modified intent to treat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Famotidine | Placebo | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (13.7) | 51.4 (12.7) | 50.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 37 | 36 | 73
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 37 | 35 | 72
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Six-minute walk distance [Mean (Standard Deviation); unit: meters] | 414 (91) | 407 (107) | 411 (99)

OUTCOME MEASURES:

1. Primary Outcome: Change in Six-minute Walk Distance
Description: To determine whether famotidine increases six-minute walk distance at 24 weeks in men and women with pulmonary arterial hypertension
Time Frame: 0 to 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Famotidine | Placebo
Number analyzed (Participants) | 40 | 39
meters | -17.0 [-43.6 to 9.7] | 4.7 [-20.1 to 29.6]

2. Secondary Outcome: Chang in Log-transformed BNP
Description: To determine whether famotidine reduces log-transformed BNP at 24 weeks
Time Frame: 0 to 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Log of pg/mL
Arm/Group | Famotidine | Placebo
Number analyzed (Participants) | 40 | 39
Log of pg/mL | -0.05 [-0.16 to 0.26] | 0.08 [-0.12 to 0.27]

3. Secondary Outcome: Proportion of Participants With New York Heart Association (NYHA) Functional Class of I or II at Week 24
Description: NYHA functional class is graded from 1 to 4 (1: no symptoms of heart failure; 2: symptoms of heart failure with moderate exertion; 3: symptoms of heart failure with mild exertion; 4: symptoms of heart failure at rest). As such, NYHA functional class 1 is considered better than NYHA functional class 4.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: Proportion participants NYHA class I/II
Arm/Group | Famotidine | Placebo
Number analyzed (Participants) | 40 | 39
Proportion participants NYHA class I/II | 0.71 [0.54 to 0.85] | 0.53 [0.36 to 0.69]

4. Secondary Outcome: Change in Right Ventricular Morphology by Echocardiogram (RV Dilation and TAPSE)
Description: To determine whether famotidine improves right ventricular morphology at 24 weeks including improved right ventricular dilation and TAPSE
Time Frame: 0 to 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: RV basal diameter (cm)/TAPSE (mm)
Arm/Group | Famotidine | Placebo
Number analyzed (Participants) | 40 | 39
RV basal diameter (cm)/TAPSE (mm)
  RV dilation | -1.5 [-3.2 to 0.3] | 0.9 [-0.9 to 2.6]
  TAPSE | 0.1 [-1.2 to 1.3] | 0.7 [-0.6 to 1.9]

5. Secondary Outcome: Change in Health Related Quality of Life (emPHasis-10 Questionnaire)
Description: To determine whether famotidine improves health related quality of life as estimated by the emPHasis-10 score (Each item on the emPHasis-10 questionnaire is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end; EmPHasis-10 scores range from 0 to 50 with higher scores indicating worse quality of life).
Time Frame: 0 to 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Famotidine | Placebo
Number analyzed (Participants) | 40 | 39
score on a scale | -1.7 [-4.2 to 0.8] | -1.3 [-3.9 to 1.2]

6. Secondary Outcome: Percent of Participants by Arm Who Added PAH Focused Care (Increased Diuretics, Escalating Doses of Pulmonary Vasodilators, and/or Adding Additional Pulmonary Vasodilators) Over 24 Weeks.
Description: To determine whether famotidine decreases the need to escalate PAH focused care (increased diuretics, escalating doses of pulmonary vasodilators, and/or adding an additional pulmonary vasodilator). The confidence interval includes a negative percent (e.g. a participant who de-escalated care).
Time Frame: 0 to 24 weeks
Measure: Number (95% Confidence Interval); unit: model-based percentage of participants
Arm/Group | Famotidine | Placebo
Number analyzed (Participants) | 40 | 39
model-based percentage of participants | 8.1 [-0.3 to 18.9] | 5.3 [-1.8 to 12.5]

7. Other Pre Specified Outcome: Invasive Hemodynamics (Sub-study): Stroke Volume Index
Description: To determine whether famotidine increases stroke volume index at 24 weeks
Time Frame: 0 to 24 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Cardiopulmonary Exercise Testing (Sub-study): Maximal Oxygen Uptake
Description: To determine whether famotidine increases maximal oxygen uptake in individuals with pulmonary arterial hypertension at 24 weeks
Time Frame: 0 to 24 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Invasive Hemodynamics (Sub-study): Hemodynamics
Description: Exploratory: To explore whether famotidine improves hemodynamics (wedge, RA, PVR) at 24 weeks
Time Frame: 0 to 24 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Cardiopulmonary Exercise Testing (Sub-study): Exercise
Description: Exploratory: To explore whether famotidine improves exercise (Ve/VCO2 ratio, total achieved wattage).
Time Frame: 0 to 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 24 weeks.
Description: Events were collected during all study visits and on a continuous basis as reported by participants or their proxies.
Arm/Group | Famotidine | Placebo
All-Cause Mortality (participants affected / at risk) | 2/40 | 1/39
Serious Adverse Events (participants affected / at risk) | 9/40 | 4/39
Other Adverse Events (participants affected / at risk) | 20/40 | 14/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Famotidine (N=40) | Placebo (N=39)
Coronavirus, Medical Device Site Infection, Metapneumovirus, Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Atrial flutter, Angina Pectoris, Cardiac Failure (Cardiac disorders) | 4 (4) | 0 (0)
syncope, encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Dehydration, Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspnea, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Famotidine (N=40) | Placebo (N=39)
Abdominal pain, dyspepsia, nausea, flatulence, discomfort (Gastrointestinal disorders) | 8 (8) | 5 (5)
Coronavirus, Influenza, Medical Device site infection, Ear infection, Metapneumovirus, Nasopharyngit (Infections and infestations) | 8 (8) | 4 (4)
Syncope, Dizziness, Headache, Dysgeusia, Encephalopathy (Nervous system disorders) | 5 (5) | 1 (1)
non-cardiac chest pain, swelling (General disorders) | 2 (2) | 0 (0)
dyspnea, hemoptysis, throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
angina, atrial flutter, cardiac failure (Cardiac disorders) | 4 (4) | 0 (0)
dehydration, hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
acute kidney injury, (Renal and urinary disorders) | 2 (2) | 0 (0)
back pain, bursitis, neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
ligament strain, muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
device malfunction (Product Issues) | 0 (0) | 1 (1)
vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03554291/Prot_001.pdf
  • Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT03554291/SAP_002.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03554291/ICF_003.pdf